CLINICAL TRIAL: NCT00946127
Title: Endoscopic Third Ventriculostomy (ETV) Versus Ventriculoperitoneal Shunting (VPS) for the Surgical Management of Normal Pressure Hydrocephalus
Brief Title: ETV Versus Shunt Surgery in Normal Pressure Hydrocephalus
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit patients and lack of efficacy in ETV arm
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Daniele Rigamonti, Professor, Johns Hopkins University
Other Study IDs: NA_00014030
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Hydrocephalus
Keywords: Normal Pressure Hydrocephalus; Communicating Hydrocephalus; Gait disorder; Cognition; Shunt; Endoscopic Third Ventriculostomy.
MeSH Terms: conditions — Hydrocephalus; Hydrocephalus, Normal Pressure; Mobility Limitation | interventions — Ventriculoperitoneal Shunt; Ventriculostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Shunt Arm: Ventriculoperitoneal Shunt
  Interventions: Procedure: Ventriculoperitoneal Shunt Placement
- ETV arm: Endoscopic Third Ventriculostomy
  Interventions: Procedure: Endoscopic Third Ventriculostomy(ETV)

INTERVENTIONS:
Procedure: Ventriculoperitoneal Shunt Placement — In the subjects who choose this arm, at the start of study- CSF (Cerebrospinal fluid ) will be shunted to peritoneum by placing a ventriculoperitoneal shunt catheter with or without shunt valves or anti-siphon device.
  Other Names: Hydrocephalus Shunt Component - Catheter-manufacturer- Medtronic Neurosurgery Inc; Codman and Hakim Shunt System--manufacturer-Codman & Shurtleff, Inc.; Medtronic PS Polyurethane Shunt--manufacturer-Medtronic Neurosurgery Inc; Miethke proGAV shunt system-manufacturer- Aesculap Inc; Medtronic PS Strata Medical Valve--manufacturer-Medtronic Neurosurgery Inc
  Groups: Shunt Arm
Procedure: Endoscopic Third Ventriculostomy(ETV) — Patients who choose to undergo ETV arm would undergo a ventriculostomy at the start of study.
  Groups: ETV arm

SUMMARY:
The purpose of this study is to test and compare the efficacy of Endoscopic Third Ventriculostomy with shunting of Cerebrospinal fluid (CSF)for treatment for patients of Normal pressure Hydrocephalus.

DETAILED DESCRIPTION:
Normal pressure Hydrocephalus is a reversible disorder of cognition and gait disorder.Currently the shunting of CSF is the recommended treatment of these patients. Even though shunts are known to be beneficial treatment of Hydrocephalus they often need treatment or revision for infection or malfunction. Endoscopic Third Ventriculostomy is a treatment without complications of shunt and is known to benefit obstructive forms of hydrocephalus.Few studies have also shown that it may be efficacious treatment Normal pressure Hydrocephalus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NPH
* Meet at least 2 of 3 Hakim and Adams diagnostic criterion for NPH (dementia, gait instability and urinary incontinence)
* Ventriculomegaly defined by CT or MRI, Evans' index > 0.3
* Clinical improvement after 3 day trial of CSF drainage.
* MMSE>24
* Informed consent from patient

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspected of Normal pressure hydrocephalus i.e. - with gait disturbances and/ or cognitive disturbances and/or urinary incontinence with dilation of ventricles on CT or MRI.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2009-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Efficacy: Cognitive outcomes using RAVLT scale. Gait Outcomes evaluated based on Tinneti Gait and Balance Test. Functional Independence evaluated using Barthel index. | 1, 3, 6, 12 months after surgery
Safety | 0 through 12 months from Surgery
  Incidence of operative complications related to insertion of a shunt or performing ETV Intra-operative hemorrhage Post Operative amnesia Post Operative hemorrhage Infections Others Incidence of complications related to either of the two procedure over long term follow-up Infection Shunt malfunction ETV closure Others

SECONDARY OUTCOMES:
Efficacy: Cognitive changes using Trails A& B. Gait changes based upon Timed Up and Go task and Gait Rite analysis. | 1 months, 3 months, 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Rigamonti, MD, FACS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Gangemi M, Maiuri F, Buonamassa S, Colella G, de Divitiis E. Endoscopic third ventriculostomy in idiopathic normal pressure hydrocephalus. Neurosurgery. 2004 Jul;55(1):129-34; discussion 134. doi: 10.1227/01.neu.0000126938.12817.dc. PMID 15214981
- [Background] Gangemi M, Maiuri F, Naddeo M, Godano U, Mascari C, Broggi G, Ferroli P. Endoscopic third ventriculostomy in idiopathic normal pressure hydrocephalus: an Italian multicenter study. Neurosurgery. 2008 Jul;63(1):62-7; discussion 67-9. doi: 10.1227/01.NEU.0000335071.37943.40. PMID 18728569
- [Background] Pujari S, Kharkar S, Metellus P, Shuck J, Williams MA, Rigamonti D. Normal pressure hydrocephalus: long-term outcome after shunt surgery. J Neurol Neurosurg Psychiatry. 2008 Nov;79(11):1282-6. doi: 10.1136/jnnp.2007.123620. Epub 2008 Mar 20. PMID 18356257
- [Background] Dusick JR, McArthur DL, Bergsneider M. Success and complication rates of endoscopic third ventriculostomy for adult hydrocephalus: a series of 108 patients. Surg Neurol. 2008 Jan;69(1):5-15. doi: 10.1016/j.surneu.2007.08.024. PMID 18054606
- [Background] Longatti PL, Fiorindi A, Martinuzzi A. Failure of endoscopic third ventriculostomy in the treatment of idiopathic normal pressure hydrocephalus. Minim Invasive Neurosurg. 2004 Dec;47(6):342-5. doi: 10.1055/s-2004-830128. PMID 15674750
- [Background] McGirt MJ, Woodworth G, Coon AL, Thomas G, Williams MA, Rigamonti D. Diagnosis, treatment, and analysis of long-term outcomes in idiopathic normal-pressure hydrocephalus. Neurosurgery. 2005 Oct;57(4):699-705; discussion 699-705. doi: 10.1093/neurosurgery/57.4.699. PMID 16239882